CLINICAL TRIAL: NCT07000552
Title: The Effect of Emotional Freedom Technique Applied to Primigravidas on Fear of Childbirth, Memory of Childbirth and Postpartum Security Sense: A Randomised Controlled Study
Brief Title: Emotional Freedom Technique During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Collaborators: EMEL EGE (Unknown)
Responsible Party: Principal Investigator, Merve Yazar, Lecturer, PhD (c), KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MerveU
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Fear of Birth; Birth Memory; Postpartum Sense of Security
Keywords: emotional freedom technique

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFT intervention (Experimental): The implementation will be carried out in accordance with EFT implementation protocols. In this context, it will be completed with 4 interviews, once a week for pregnant women. i Each EFT session will last 15 minutes.
  Interventions: Other: EFT intervention
- Control grup (No Intervention): There will be no intervention. Women in the intervention groups will be followed up for 4 weeks and will receive standardised care. The final test will be administered in the postnatal period

INTERVENTIONS:
Other: EFT intervention — The intervention groups will be followed up for 4 weeks and 4 EFT therapies will be applied, one session per week.
  Arms: EFT intervention

SUMMARY:
Emotional Freedom Technique (EFT), also known as "Tapping Therapy" and "Needleless Acupuncture", is a new and emerging complementary and energy-based therapy. It is a psychophysiological intervention combining cognitive behavioural therapy, exposure therapy and physical stimulation using acupressure points. This research will be conducted to evaluate the effect of emotional liberation technique applied to primigravidas on fear of childbirth, birth memory and postpartum feelings of safety. The research will be conducted between January 2025 and October 2025 in Konya Necmettin Erbakan University Faculty of Medicine Hospital, Department of Obstetrics and Gynaecology, Pregnant Outpatient Clinic with primiparous women planning vaginal delivery. This research is planned to be conducted with two groups, EFT intervention and control group. The population of the study consisted of pregnant women who applied to the pregnancy outpatient clinic of a university hospital located in the city centre of Konya province and were evaluated for eligibility.

ELIGIBILITY:
Inclusion Criteria:

* Primary education level or higher
* Able to speak, understand and write Turkish,
* 18 years of age or older,
* Residing in Konya province,
* No disability for vaginal delivery,
* Primigravida,
* Anxiety level of 1 or higher when measured with the subjective discomfort unit scale,
* Pregnant women who are at 32 weeks of gestation or above according to the last menstrual date or according to calculations made with USG data for pregnant women who do not know the last menstrual date.

Exclusion Criteria:

* Pregnant individuals with high-risk pregnancies,
* Those who have undergone infertility treatment,
* Those with any fetal health problems,
* Those with physical or mental illnesses,
* Those with a cesarean section indication or who plan to deliver via cesarean section,
* Those with chronic and/or psychiatric health issues and those who have participated in any childbirth preparation education were excluded from the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
EFT Intervention | 4 weeks
  Women with a gestational age of 32 and above will be administered the Subjective Experience Unit scale before and after the intervention. The Subjective Experience Unit scale was developed by Hartmann with the "Events Psychology" approach in order to measure the energy flow in the energy body. This scale is used to determine the emotional intensity of the person at the beginning and at the end of the EFT session. In this scale, scoring is made between -10 and +10. -10 is the greatest pain, disappointment, fear, stress, sadness or discomfort imaginable, while +10 is the highest level of joy, happiness or feeling great.
  The final tests will be administered in the postnatal period. In the postnatal period, Wijma Birth Anticipation/Experience Scale, Birth Memory and Recall Scale, Postnatal Feelings of Security Scale and Postnatal Interview Form were completed.
Control grup | 4 week
  Pregnant women in the control group will be called once a week and asked to score the SUE scale and recorded, and 1 hour later, they will be asked to score the SUE scale again without any intervention. Final tests will be administered in the postnatal period.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No